CLINICAL TRIAL: NCT06951009
Title: Establishing Baseline Sysmex UF-5000 Flow Cytometer Results in Healthy Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Stephen J. Jordan, Principal Investigator, Indiana University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 26774
Record Dates: First submitted 2025-04-12; First posted 2025-04-30 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-06

CONDITIONS: Urethritis; Healthy Men Age 18-50 With no Urethral Symptoms
MeSH Terms: conditions — Urethritis | interventions — Urinalysis

STUDY DESIGN:
Intervention Model Description: Participants with an odd birth year will use the Colli-Pee during the first week; even birth year participants will use the Colli-Pee during the second week.
  Participants with an odd birth year will use the standard-of-care 60 mL urine cup during the second week; even birth year participants will use the urine cup during the first week.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Colli-Pee collection followed by standard-of-care urine collection cup (Active Comparator): Participants with an odd birth year will collect urine using the Colli-Pee device during Week 1 and with the standard-of care urine cup during Week 2.
  Interventions: Device: Colli-Pee; Device: standard of care 60 mL urine cup; Diagnostic Test: Urinalysis; Diagnostic Test: Sysmex UP-5000
- Standard-of-care urine collection followed by Colli-Pee collection (Active Comparator): Participants with an even birth year will collect urine using the standard-of-care urine cup during Week 1 and with the Colli-Pee device during Week 2.
  Interventions: Device: Colli-Pee; Device: standard of care 60 mL urine cup; Diagnostic Test: Urinalysis; Diagnostic Test: Sysmex UP-5000

INTERVENTIONS:
Device: Colli-Pee — The Colli-Pee device is a first void urine self-sampling device. Participants will collect urine samples with this device three times during one week of study participation. Urine sample collection with this device will occur either in Week 1 or Week 2 of study participation, depending on the Participant's Arm assignment.
Device: standard of care 60 mL urine cup — Participants will collect clean catch urine samples with this device three times during one week of study participation. Urine sample collection with this device will occur either in Week 1 or Week 2 of study participation, depending on the Participant's Arm assignment.
Diagnostic Test: Urinalysis — Participant samples will be analyzed by urinalysis to evaluate for leukocyte esterase (LE).
Diagnostic Test: Sysmex UP-5000 — Participant samples will be analyzed by the Sysmex UP-5000 to evaluate for white blood cells (WBCs) per microliter.

SUMMARY:
Acute urethritis (inflammation of the male urethra) affects millions of men in the United States each year.

Effective management of STIs is complicated by asymptomatic infections, as men often delay seeking care until symptoms become severe. Yet, even men without symptoms can show measurable evidence of urethritis. Therefore, a cheap, simple, and non-invasive point-of-care (POC) test, providing results within 30 minutes, could significantly enhance STI management by facilitating early diagnosis and treatment.

A new diagnostic method, urine flow cytometry, has shown potential in hospital settings for accurately detecting inflammation by counting white blood cells (infection-fighting cells) in urine samples. The Sysmex UF-5000 flow cytometer, a state-of-the-art device, may offer a non-invasive, cost-effective, and accurate method to diagnose urethritis compared to traditional Gram stains and urinalysis, potentially extending its use beyond specialized clinics.

This study aims to determine the efficacy and precision of the Sysmex UF-5000 analyzer in diagnosing urethritis using first-catch urine samples. Additionally, the study seeks to evaluate whether urine collected using the 10 mL Colli-Pee device provides greater accuracy and precision compared to the standard urine cup (30-60 mL) when used with urine flow cytometry and LE urinalysis.

DETAILED DESCRIPTION:
Acute urethritis (i.e., inflammation of the male urethra) affects millions of men within the United States annually. In young sexually active men, urethritis is most commonly caused by the sexually transmitted infections (STI) Neisseria gonorrhoeae (GC, causes gonorrhea) and Chlamydia trachomatis (CT, causes chlamydia), but can also be caused by a lengthening list of known and emerging pathogens that cause "nongonococcal urethritis" (NGU). STI management has proven challenging due to the prevalence of asymptomatic infections and because men often fail to seek STI care until they experience pronounced symptoms. However, even without urethral symptoms, most men with a urethral STI have measurable evidence of urethritis. Thus, a cheap, simple, and non-invasive point of care (POC) test (i.e., results available within 30 minutes) that accurately detects urethritis could be a game changer in STI management as asymptomatic infections could be detected and treated, potentially decreasing the risk of spreading STIs to sexual partners.

Currently, the only widely used POC test available for diagnosis of urethritis in men in the US is Gram stain microscopy of a urethral swab smear. This approach has been shown to be highly effective for identifying men who have urethritis and has 95% sensitivity for diagnosing GC in symptomatic men [4]. Although the urethral swab remains the gold standard test to diagnose urethritis at the POC, it is rarely used outside of specialized STI clinics given its many limitations, which include: (1) it often elicits severe pain, and in rare cases can permanently damage the urethra; (2) it requires specialized instrumentation (an inverted microscope with a 1000x objective) and Gram stain reagents; (3) it must also be administered and interpreted by trained personnel that have different inter-operator accuracy in reporting results, and (4) anxiety associated with this procedure is a common reason men cite for delaying STI care and failing to return for follow-up visits. In many other clinical settings, POC screening for STIs would be highly desirable, for example during annual wellness exams of high-risk male adolescents; screening with specific STI nucleic acid amplification tests (NAATs) is not cost-effective in low-risk populations and the urethral swab procedure is unacceptable in these populations. As an alternative approach, a few investigators have evaluated Leukocyte esterase (LE) testing as part of a routine urinalysis using first-catch urine to diagnose urethritis, but the low sensitivity and specificity of this approach has limited its use to resource-limited settings.

Flow cytometry is routinely used in clinical settings to identify populations of cells (e.g., neutrophils, red blood cells for whole blood counts) from blood and urine. Modern flow cytometers are highly automated, rapid, and inexpensive to run, which makes them an optimal assay for screening for urethritis by detecting elevated neutrophils in asymptomatic men. Interestingly, several recent publications have shown that flow cytometric analysis of urine can be used to diagnose urethritis with comparable sensitivity and specificity to the urethral Gram stain smear. However, most of these studies did not use state-of-the-art flow cytometers, did not calibrate Gram stain to flow cytometric results directly, and did not diagnose the sensitivity/specificity of this approach for detection of a broad section of urethral STI. The investigators hypothesize that the state-of-the-art flow cytometer analyzer, Sysmex UF-5000, may be able to similarly provide a non-invasive and cost-effective approach for urethritis diagnosis in men using first-catch urine when compared to Gram stain and urinalysis. A prior version, the Sysmex UF-1000i, has been shown to be promising in detection of urinary tract infections, but has not yet been studied in STIs. The UF-5000 could be a powerful screening approach for urethral STI that could be employed in a broad range of clinical settings, not just specialized STI clinics. Separately, if urine flow cytometry could be optimized to yield similar sensitivity to the Gram stain smear, the investigators suspect this approach would rapidly replace the Gram stain smear in clinical practice which in turn would improve patient capture and retention.

The investigators will recruit healthy men aged 18 to 50 who, after consenting to participate, will be assigned to start collecting a urine specimen three times week (typically, Monday, Wednesday, and Friday) for two weeks.

The device used to collect urine will be either a Colli-Pee or a standard-of-care 60 ml sterile urine cup. Participants with an odd birth year will use the Colli-Pee during the first week; even birth year participants will use the Colli-Pee during the second week.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 18 to 50.
* No urethral symptoms (discharge, dysuria)

Exclusion Criteria:

* History of genital surgery or known urethral abnormalities
* Testing positive for gonorrhea and chlamydia
* Diagnosis of a sexually transmitted infection within the last year.
* Not available to collect a urine specimen in the morning 3x/week for 2 weeks

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — assigned male at birth
Enrollment: 20 (Actual)
Dates: Start 2025-04-09 (Actual); Primary Completion 2025-05-07 (Actual); Study Completion 2025-05-07 (Actual)

PRIMARY OUTCOMES:
Detection of white blood cells in single sample | Three days during Week 1 and three days during Week 2
  Participants will provide urine samples on three days during each week of participation, for a total of 2 weeks. Urine samples collected in standard of care urine cups and Colli-Pee devices will be compared for white blood cells (WBC) per microliter, as detected by the Sysmex UP-5000. The UF5000 results will be the continuous variable of "WBCs per microliter" of urine.
Detection of leukocyte esterase (LE) in single sample | Three days during Week 1 and three days during Week 2
  Participants will provide urine samples on three days during each week of participation, for a total of 2 weeks. Urine samples collected in standard of care urine cups and Colli-Pee devices will be compared for leukocyte esterase as detected by urinalysis. For the urinalysis, the categorical results will be "neg", "1+", "2+", "3+", and "4+" leukocyte esterase.
Detection of white blood cells in repeat sampling | Three days during Week 1 and three days during Week 2
  Participants will provide urine samples on three days during each week of participation, for a total of 2 weeks. Urine samples collected in standard of care urine cups and Colli-Pee devices will be compared for white blood cells (WBC) per microliter, as detected by the Sysmex UP-5000. The UF5000 results will be the continuous variable of "WBCs per microliter" of urine. The average of 3 sample collections will be evaluated.
Detection of leukocyte esterase (LE) in repeat sampling | Three days during Week 1 and three days during Week 2
  Participants will provide urine samples on three days during each week of participation, for a total of 2 weeks. Urine samples collected in standard of care urine cups and Colli-Pee devices will be compared for leukocyte esterase as detected by urinalysis. For the urinalysis, the categorical results will be "neg", "1+", "2+", "3+", and "4+" leukocyte esterase. The average of 3 sample collections will be evaluated.
Detection of white blood cells over time | Three days during Week 1 and three days during Week 2
  Participants will provide urine samples on three days during each week of participation, for a total of 2 weeks. Urine samples collected in standard of care urine cups and Colli-Pee devices will be compared for white blood cells (WBC) per microliter, as detected by the Sysmex UP-5000. The UF5000 results will be the continuous variable of "WBCs per microliter" of urine. Specimens will be compared at 0 hours, 1 hour, 2 hours, 4 hours and 8 hours.
Detection of leukocyte esterase (LE) over time | Three days during Week 1 and three days during Week 2
  Participants will provide urine samples on three days during each week of participation, for a total of 2 weeks. Urine samples collected in standard of care urine cups and Colli-Pee devices will be compared for leukocyte esterase as detected by urinalysis. For the urinalysis, the categorical results will be "neg", "1+", "2+", "3+", and "4+" leukocyte esterase. Specimens will be compared at 0 hours, 1 hour, 2 hours, 4 hours and 8 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Jordan, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
Information and specimens collected for this study may be used for other research studies or shared with other researchers who are conducting their own research studies. This may include sharing with researchers outside Indiana University and sharing with private companies. It may also include making the information available in public and private databases of research data so that other researchers can use the information to answer research questions.
  If study staff share information or specimens in this way, they will remove information that could identify the subject(s), such as name and contact information, before any information or specimens are shared.
  Due to privacy concerns, IPD will not be shared.